CLINICAL TRIAL: NCT04026243
Title: Ultrasound-Guided Transversalis Fascia Plane Block Versus Transmuscular Quadratus Lumborum Block for Post-operative Analgesia in Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hany Mohammed El-Hadi Shoukat Mohammed, lecturer of anesthesia, pain management and SICU, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-48-2018
Record Dates: First submitted 2019-07-15; First posted 2019-07-19 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Pain Management of Inguinal Herniorrhaphy
Keywords: ultrasound guided regional blocks; Transversalis Fascia Plane Block; Quadratus Lumborum Block; inguinal herniorrhaphy; Pain management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL group (n = 25) (Active Comparator): After general anesthesia (GA), patient will be placed in lateral position with side to be anesthetised upwards. U/S probe will be placed in the transverse plane at the abdominal flank immediately cranial to the iliac crest. Then moved dorsally until the QL muscle is identified with its attachment to lateral edge of the transverse process of the L4 vertebral body with identification of shamrock sign. The needle is inserted in-plane to transducer (lateral edge) and tip of needle is advanced through the QL muscle. Once the tip of the needle correctly placed and confirmed by negative aspiration, 2 ml of normal saline will be instilled to confirm correct separation of the plane. Following this, 30 ml of 0.25% bupivacaine will be injected between the QL and psoas major.
  Interventions: Procedure: QL block
- TF group (n = 25) (Active Comparator): After GA, patient will be placed in lateral position with side to be anesthetised upwards. U/S probe will be placed in midaxillary line just cephalad to the iliac crest. Scanning anteriorly will identify the three muscles of the anterior abdominal wall. The transversus abdominis typically tapers to form a hyper echoic aponeurosis that passes posterior to quadratus lumborum. Scan will be continued posteriorly to visualize solid organs or viscera deep to the transversus abdominis. The needle will be positioned such that it enters the skin anterior to the ultrasound probe and passes in-plane posterolateral through the three lateral abdominal muscles. Once the tip of the needle correctly placed and confirmed by negative aspiration, 2 ml of normal saline will be instilled to confirm correct separation of the plane. Following this, 30 ml of 0.25% bupivacaine will be injected between the transversus abdominis muscle and the transversalis fascia anterolateral to quadratus lumborum.
  Interventions: Procedure: TF block

INTERVENTIONS:
Procedure: QL block — U/S guided Transmuscular Quadratus Lumborum Block
  Arms: QL group (n = 25)
Procedure: TF block — U/S guided Transversalis Fascia Plane Block
  Other Names: TFP block
  Arms: TF group (n = 25)

SUMMARY:
Regional blocks as a part of multimodal analgesia can improve pain control in the postoperative period. The transversalis fascia plane (TFP) block can block the proximal portions of the T12 and L1 nerves, while the main advantage of the Quadratus Lumborum (QL) block is the possible extension of the local anesthetic beyond the transversus abdominis plane (TAP) plane spreading into the thoracic paravertebral space and anesthetizing both the lateral and anterior cutaneous branches from T7 to L1. the aim of this study is to compare effectiveness of ultrasound-guided transversalis fascia plane block to trans-muscular quadratus lumborum block in providing postoperative analgesia in patients undergoing unilateral inguinal hernia repair.

DETAILED DESCRIPTION:
This prospective randomized controlled study will include 50 patients (25 in each group) of American Society of Anesthesiologist (ASA) I and II physical status who will undergo unilateral inguinal herniorrhaphy under general anesthesia. The investigators hypothesize that ultrasound-guided trans-muscular quadratus lumborum block will be more effective than ultrasound guided transversalis fascia plane block in providing postoperative analgesia in these type of patients. Randomization will be done by a computer-generated random numbers. Patients will be blinded to the study groups. All patients will undergo a thorough pre anesthetic check-up and will be premedicated with metoclopramide 10 mg intravenously.

In the operation theatre, an 18-gauge intravenous (IV) catheter will be placed and monitoring devices will be attached which will include electrocardiograph (ECG) using (GE-Datex Ohmeda 5 lead ECG cable), pulse oximetry (SpO2) using (GE- Datex Ohmeda adult finger spO2 sensor), non-invasive blood pressure (NIBP) using (GE-Datex Ohmeda NIBP cuff, adult double tube with bag). Emergency drugs and equipment will be ready and prepared. Numeric pain rating scale will be explained clearly to all patients before conduction of anesthesia.

Anesthesia will be induced with fentanyl (2 mcg/kg) and propofol (1.5-2.5 mg/kg) and atracurium besylate (0.5 mg/Kg). An endotracheal tube will be inserted, and controlled ventilation will be adjusted to maintain normocapnia. Anesthesia will be maintained with sevoflurane at 1% and boluses of atracurium (0.1 mg/Kg) every 30 min. All patients will be given 1 g intravenous paracetamol, together with 4 mg ondansetron 10 min prior to the end of surgery for postoperative nausea and vomiting prophylaxis.

The patients will be classified into two equal groups; Group QL (n=25) and group TF (n=25).

All blocks will be performed on patients, following general anesthesia induction and endotracheal tube insertion, under guidance of a digital ultrasonic diagnostic imaging system (Mindray®, china), using a low frequency (2-6 MHz) curvilinear probe and a 100-150-mm short-bevel echogenic needle. Before ultrasound scanning, the operator will wear sterilized gown and gloves following routine scrubbing, flank skin will be prepared by antiseptic solution and fenestrated drape and dressings will be used for all procedures. After surgical disinfection of ipsilateral flank and protection of the ultrasound probe with a sterile ultrasound probe cover, sterile gel will be applied prior to scanning.

After skin closure, inhalational anesthesia will be discontinued and reversal of muscle relaxation with atropine (0.02 mg/Kg) and neostigmine (0.05 mg/Kg) will be administered IV after return of patient's spontaneous breathing. Patient will then be transferred to post anesthesia care unit (PACU) for complete recovery and monitoring.

In the PACU; rescue analgesia in the form of intravenous nalbuphine (in 5 mg increments) will be given for a numerical pain score more than 4 in the immediate postoperative period.

The block will be considered a failed block if the patient required more than one 5mg dose of nalbuphine in the first hour postoperatively.

In the ward; rescue analgesia will be given in the form of intravenous nalbuphine (in 5 mg increments) and repeated if needed every half an hour with a maximal dose of 60 mg in 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients of ASA classification grade I and II,
* aged above 18 years old and less than 65 years old,
* of both sexes,
* body mass index (BMI) below 35,
* who had a capacity to rate pain on a numeric rating scale (NRS) of 0 to --underwent non-recurrent unilateral inguinal hernia repair

Exclusion Criteria:

* patient refusal
* patient aged < 18 or > 65 years old,
* ASA classification > II, BMI < 35
* those with previous difficulty in evaluating their level of pain
* any contraindications for local anesthesia as: patient refusal of local anesthesia injection, coagulopathy( defined as either thrombocytopenia (platelet count below 100,000 platelets per microliter and/or prothrombin time greater than 14 seconds ), therapeutic anticoagulation, presence of skin infection or hematoma in the vicinity of the puncture site or those with known allergy to any of the study drugs

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
postoperative numeric pain rating scale (NRS) from 0 to 10 | Measured at 30 minutes postoperatively.
  Patient-assessed resting and movement-induced pain on a numeric pain rating scale of 0 to 10 (higher score will be taken).

SECONDARY OUTCOMES:
postoperative numeric pain rating scale (NRS) from 0 to 10 | Measurements at 10 minutes, 30 minutes, 60 minutes and 90 minutes after surgery, and at 24 hours postoperatively
  Patient-assessed resting and movement-induced pain on a numeric pain rating scale of 0 to 10 (higher score will be taken).
number of increments of rescue analgesia | from 30 mintes up to 24 hours postoperative
  number of increments of nalbuphine needed in the immediate postoperative period up to 24 hours postoperative
level of sensory block in the immediate postoperative period | 10 minutes after PACU admission
  determined by application of a cold, wet cotton swab: anesthesiologist will compare reaction to the stimulus between the nerve territories on the surgery side to the contralateral territory. Sensitivity will be graded on a scale of 0 to 2 (2: normal sensitivity to cold; 1: hypoesthesia; and 0: anesthesia)
Easiness of performance of the block | once during block performance
  operator will be asked and his answer will be rated on a simple verbal scale (easy/moderately difficult/difficult) and defined as follows:Easy block: if successful block after the 1st skin puncture and no need for needle image optimization (no adjustment of depth, gain, or focus to visualize the needle path). Moderately difficult block: if successful block after more than one skin puncture attempt or with the need for needle image optimization (as adjustment of depth, gain, or focus to visualize the needle path).Difficult block: if successful block after > one skin puncture attempt and with the need for needle image optimization (as adjustment of depth, gain, or focus to visualize the needle path). N.B: successful block means adequate hydrodissection under U/S
Block performance time in minutes | from U/S probe contact with skin till needle withdrawal up to 30 minuteas afteintubation
  Block performance time in minutes (defined as time from probe contact with skin till needle withdrawal
Patient satisfaction regarding pain management | rated 6 hours after surgery
  a verbal questionnaire (how did you find your pain sensation in the past 6 hours?), patient will describe his/her satisfaction regarding pain management as being (very satisfied, satisfied, not very satisfied, dissatisfied),
incidence of adverse effects, | postoperative up to 24 hours
  incidence of adverse effects, such as postoperative nausea and vomiting, urinary retention, and local anesthetic toxicity
Failure rate of the block | in the first hour postoperatively
  the block will be considered a failed block if when the patient required more than two 5 mg doses of nalbuphine in the first hour postoperatively

OTHER OUTCOMES:
heart rate (HR) | up to 60 minutes after removal of endotracheal tube
  in beat per minute,1 minute before induction of anesthesia (T0), 5 minutes after induction of anesthesia (T1), 5 minutes after injection of local anesthesia (LA) (T2) performing the block, 15 minutes after injection of LA (T3), 30 minutes after injection of LA (T4), 45 minutes after injection of LA (T5), 5 minutes after removal of endotracheal tube (T6), 15 mintes after removal of endotracheal tube (T7), 30 minutes after removal of endotracheal tube (T8), and 60 minutes after removal of endotracheal tube (T9).
systolic blood pressure (SBP) | up to 60 minutes after removal of endotracheal tube
  in mmHg,1 minute before induction of anesthesia (T0), 5 minutes after induction of anesthesia (T1), 5 mintes after injection of LA (T2) performing the block, 15 minutes after injection of LA (T3), 30 minutes after injection of LA (T4), 45 minutes after injection of LA (T5), 5 minutes after removal of endotracheal tube (T6), 15 minutes after removal of endotracheal tube (T7), 30 minutes after removal of endotracheal tube (T8), and 60 minutes after removal of endotracheal tube (T9).
mean arterial blood pressure (MAP) | up to 60 minutes after removal of endotracheal tube
  in mmHg, 1 minute before induction of anesthesia (T0), 5 minutes after induction of anesthesia (T1), 5 mintes after injection of LA (T2) performing the block, 15 minutes after injection of LA (T3), 30 minutes after injection of LA (T4), 45 minutes after injection of LA (T5), 5 minutes after removal of endotracheal tube (T6), 15 minutes after removal of endotracheal tube (T7), 30 minutes after removal of endotracheal tube (T8), and 60 minutes after removal of endotracheal tube (T9).
Duration of surgery | time from skin incision till skin closure up to 180 minutes after GA induction
  in minutes
Duration of general anesthesia | time from induction of GA till removal of endotracheal tube up to 18 minutes after GA induction
  in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Hany MES Mohammed, MD, Principal Investigator — www.kasralainy.cu.edu.eg
Locations (1):
- Hany Mohammed El-Hadi Shoukat Mohammed, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol